CLINICAL TRIAL: NCT05723627
Title: Comparison of Remimazolam and Propofol Effect on Oxygenation Reservoir During Diagnostic Gastric Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2022-1369
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Diagnostic Gastric Endoscopy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Patient group who receives remimazolam for sedation during endoscopy
  Interventions: Drug: Remimazolam besylate
- Propofol (Active Comparator): Patient group who receives propofol for sedation during endoscopy
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam besylate — Patients in this group receives 0.1mg/kg of remimazolam to induce sedation prior to endoscope insertion.
  Arms: Remimazolam
Drug: Propofol — Patients in this group receives 0.5mg/kg of propofol to induce sedation prior to endoscope insertion.
  Arms: Propofol

SUMMARY:
Propofol is one of the most commonly used sedative in endoscopic procedures, while its potency to induce respiratory depression may threaten patient safety. Remimazolam is known to less likely induce hemodynamic instability when compared to propofol, yet its favorable effects are not clearly evaluated in endoscopic procedures. Hence, this study aimed to compare hemodynamic effects of remimazolam and propofol, by evaluating oxygen reserve index (ORI) in patients scheduled for diagnostic gastric endoscopy.

ELIGIBILITY:
Inclusion Criteria:

Patients (age 19~80 yrs, ASA Class I~III, ECOG 0~1) who are scheduled for elective diagnostic gastric endoscopy

Exclusion Criteria:

Pregnancy Allergy to remimazolam or propofol Underlying pulmonary diseases or obstructive sleep apnea Hypotension (SBP <80mmHg) or hypoxemia (SpO2 <90%) assessed prior to procedure

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Incidence of Oxygen Reserve Index (ORI) drop to 0.00 during sedation | Evaluation begins after sedative administration until the end of endoscopic procedure.
  Incidence of Oxygen Reserve Index (ORI) drop to 0.00 will be evaluated after sedative administration, until the end of endoscopic procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Kwan Shin, Principal Investigator — Department of Internal Medicine, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea